CLINICAL TRIAL: NCT02225561
Title: SNPeCPR Pour la prIse en Charge Des Arrêts CaRdiaques Extrahospitaliers
Brief Title: SNPeCPR In Cardiac Arrest REsuscitation
Acronym: SICARE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinuation of the experimental treatment being tested
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P130946; 2014-002010-24 (EudraCT Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Cardiopulmonary Arrest
Keywords: Cardiopulmonary resuscitation; Nitroprusside; Transthoracic; Impedances
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): Pharmaco- mechanical optimization
  Interventions: Procedure: pharmaco- mechanical optimization
- Mechanical optimization only (Active Comparator): Mechanical optimization only
  Interventions: Procedure: mechanical optimization only

INTERVENTIONS:
Procedure: pharmaco- mechanical optimization — Getting started as soon as possible cardiopulmonary resuscitation (CPR) mechanical ( LUCAS 2) with inspiratory impedance valve ( ResQPOD ) performed according to the 2015 recommendations of the European Resuscitation Council . It will be carried out continuously without a break for control pulse until the first defibrillation attempt.
  As soon the peripheral intravenous or intraosseous line is set the intervention group will receive an injection of 2 mg of sodium nitroprusside. 4 minutes after the first injection, a second and last injection of 1 mg of sodium nitroprusside will be realized.- The preparation procedure of the sodium nitroprusside will be:
  * Using a "pomping needle" and the provided syringe 4 ml of the solvent (Water for Injections, WFI) will be take.
  * The 4 ml of WFI will be empty in the 50 mg vial of lyophilisate sodium nitroprusside to solubilize the product.
  * Always with the needle and 20 ml syringe, the 4 ml of this solution (50 mg in 4 ml) will be collect.
  Arms: Intervention arm
Procedure: mechanical optimization only — Getting started as soon as possible cardiopulmonary resuscitation (CPR) mechanical ( LUCAS 2) with inspiratory impedance valve ( ResQPOD ) performed according to the 2015 recommendations of the European Resuscitation Council . It will be carried out continuously without a break for control pulse until the first defibrillation attempt.
  Arms: Mechanical optimization only

SUMMARY:
Approximately 50,000 patients are victims of out of hospital cardiac arrest every year in France. Despite cardiopulmonary resuscitation (CPR) and many studies on the topic resuscitation survival after cardiac arrest remains low (1-8%) and has not changed significantly over the past five decades.It has recently been shown that the combination of different non-invasive therapies, cardiopulmonary resuscitation with mechanical CPR with automated compression / decompression and an impedance threshold device, can increase the rate of return of spontaneous circulation and short and long term survival after cardiac arrest.We propose to study a new cardiopulmonary resuscitation called SNPeCPR (Sodium nitroprusside enhanced cardiopulmonary resuscitation), which includes two components:a) a mechanical component: cardiopulmonary resuscitation with automated mechanical external chest compression and an impedance threshold deviceb) a pharmacological component: sodium nitroprusside, an effective arterial vasodilator that decrease vascular resistance, and improve flow in vital organs.Our hypothesis is that SNPeCPR should improve the return of spontaneous circulation rate during cardiac arrest.

DETAILED DESCRIPTION:
1. OBJECTIVES The objective of this study is to demonstrate the superiority of Sodium nitroprusside enhanced cardiopulmonary resuscitation (SNPeCPR) on optimized standard cardiopulmonary resuscitation.

   SNPeCPR includes two components:
   1. a mechanical component: cardiopulmonary resuscitation with automated mechanical external chest compression and an impedance threshold device
   2. a pharmacological component: sodium nitroprusside, an effective arterial vasodilator that decreasing vascular resistance, facilitates flow elevation in vital organs.

   1.1. Main Objective : Assess the interests of the administration of sodium nitroprusside during enhanced cardiopulmonary resuscitation.

   1.2. Secondary Objectives : To evaluate the effect of sodium nitroprusside on various parameters before and after the return of spontaneous circulation.

   1.3. Outcome Measures : In this declaration, all the criterions measures before ROSC have been note as t=0 minute.

   For the elements were the timeframe is a variable, ICU and hospital discharge, they have been declare at 1 and 2 weeks respectively.
2. NAME AND DESCRIPTION OF THE INVESTIGATIONAL DRUG Sodium nitroprusside (SNP) is a potent vasodilator that we will use in cardiac arrest to optimize vital organs perfusion. The purpose of CPR is to provide oxygenated blood to vital organs that are most susceptible to ischemic insult (brain and heart). Since the mechanical combination (cardiopulmonary resuscitation with automated mechanical external chest compression and an impedance threshold device) provides excellent perfusion pressure, the flow should be optimized pharmacological with vasodilation. The SNP reduces arterial vasoconstriction and enhances microcirculation. Furthermore, SNP significantly reduces vascular resistance and decreases cardiac ejection afterload. Therefore, SNPeCPR can significantly increase the flow of blood and optimize carotid and coronary flow.
3. PROCEDURE During cardiac arrest resuscitation, patients will be included in the study after the investigator has verified the inclusion and non-inclusion criterion. A sealed box containing SNP or the placebo will then be open in the increasing numbers of randomization list.

   Whatever the allocated treatment (nitroprusside or Placebo [5% glucose solution]), cardiopulmonary resuscitation protocol will be realize as recommended by the 2010 European Resuscitation Council and described as follows:
   * cardiopulmonary resuscitation will be performed continuously without posing for control pulse until the first defibrillation attempt. As soon as possible manual CPR will be replace by automated mechanical external chest compression (LUCAS® - Lund University Cardiopulmonary Assist System) and an impedance threshold device (ResQPOD®).
   * placement of a peripheral intravenous (IV) or intraosseous (IO) line. This placement will be privileged to intubation,
   * when the peripheral intravenous or intraosseous line is set, 1.96 mg sodium nitroprusside (SNP) / placebo will be injected, followed by injection of 10 ml saline for intravenous flush (t = 0 minutes).
   * 1 mg of epinephrine will be injected at t = 2 minutes,
   * an external electric shock (EEC) will be realized at t = 3 minutes when the electric heart type allows it (ventricular fibrillation or ventricular tachycardia),
   * 0.98 mg sodium nitroprusside / placebo will be injected at t = 4 minutes, followed by an injection of 10 ml of saline for intravenous flush.
   * 1 mg adrenaline will be injected at t = 7 minutes, the injection will be repeated every 5 minutes until return of spontaneous circulation or ending of the resuscitation decided by the emergency physician.
   * an external electric shock (EEC) will be realized at t = 6 minutes when the electric heart type allows, then external shock will be repeated every 3 minutes until return of spontaneous circulation or ending of the resuscitation decided by the emergency physician.

   During that resuscitation the following parameters will be collected:
   * The type of cardiac arrest (place of cardiac arrest [home, public place, stadium …], cardiac arrest before a witness or prompt rescue team, cardiac massage by the witness or prompt rescue team, durations between collapse and the start of resuscitation, non-specialized / specialized resuscitation, defibrillation shock by the witness or prompt rescue team), ETCO2, blood pressure and SpO2.
   * the initial electrical rhythm (defined by ECG) by the mobile intensive care unit (MICI) and ECG 5 minutes after return of spontaneous circulation.
   * arterial blood gas lactate
   * troponin (24 hours after ROSC)
   * liver function (24 hours after ROSC)
   * creatinine (24 hours after ROSC)
   * echocardiography (4 and 24 hours after ROSC)
4. EXPECTED DURATION OF PARTICIPATION OF PEOPLE AND DESCRIPTION OF THE TIMING AND DURATION OF THE RESEARCH.

   Duration of intervention: 4 minutes Inclusion time: 30 months duration of participation (+ monitoring treatment): 6 months Total duration of the study: 3 years
5. RANDOMIZATION Randomization will be realized by block and will be stratified by center. The boxes are numbered and contain drugs specified by the randomization arm. Randomization will be done by assigning at each inclusion a box taken in order of increasing numbers of the randomization list. The randomization list will be established under the responsibility of the clinical research unit.
6. MONITORING COMMITTEE A monitoring committee will conduct an interim analysis after the inclusion of 50% and 75% of patients and will decide to stop or continue the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with out of hospital cardiac arrest
* Age> 18 years and <75 years
* Initial Rhythm: Ventricular fibrillation or ventricular tachycardia or pulseless electrical activity

Exclusion Criteria:

* out of hospital cardiac arrest of non-cardiac origin:

  * trauma
  * anoxic, including drowning
  * hemorrhage,
  * overdose (drugs),
  * drug,
  * electric
* Do Not Resuscitate Order,
* obvious signs of clinical death (decomposition, cadaveric rigidity, decapitation)
* recent sternotomy (<6 months or recent scar)
* Contraindications related to sodium nitroprusside

  * Women of childbearing age (between 18 and 55 years)
  * Other contra-indications will usually not known during resuscitation in case of presence of a relative rescue team must be searched: Hypothyroidism, Sulfuryl transferase deficiency (rhodanese Lang) currently recognized in patients with Leber optic atrophy, tobacco amblyopia or severe hepatic impairment.
* Obesity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Rate of return of spontaneous circulation (ROSC) | at 5 minutes
  Rate of return of spontaneous circulation (ROSC) defined as a central pulse (carotid or femoral) palpable for more than 5 minutes

SECONDARY OUTCOMES:
ETCO2 | at 0, 5 and 60 minutes
  ETCO2 (before ROSC, 5 and 60 min after ROSC)
Blood pressure | at 5 and 60 min
  at 5 and 60 min after ROSC
ECG | at 0, 5 and 60 minutes
  ECG (before ROSC, 5 min after ROSC)
SpO2 | at 0, 5 and 60 minutes
  SpO2 (before ROSC, 5 and 60 min after ROSC)
Arterial blood gases with lactate | at 0 and 5 minutes; 1, 4 and 24 hours
  arterial blood gases with lactate (before ROSC, 5 min, 1, 4 and 24 hours after ROSC)
Troponin | at 24 hours
  troponin (24 hours after ROSC)
Liver function | at 24 hours
  liver function (24 hours after ROSC)
Creatinine | at 24 hours
  creatinine (24 hours after ROSC)
Echocardiography | at 4 and 24 hours
  echocardiography (4 and 24 hours after ROSC)
Survival | 1, 4 and 24 hours, 1 week, 2 weeks, 1 and 6 months
  survival (1, 4 and 24 hours after ROSC, ICU and hospital discharge, 1 and 6 months)
Neurological score | 1 week, 2 weeks, 1 and 6 months
  neurological score (ICU and hospital discharge, 1 and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PLAISANCE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SMUR - Hôpital Lariboisière, Paris, France

REFERENCES:
- [Background] Schultz J, Segal N, Kolbeck J, Caldwell E, Thorsgard M, McKnite S, Aufderheide TP, Lurie KG, Yannopoulos D. Sodium nitroprusside enhanced cardiopulmonary resuscitation prevents post-resuscitation left ventricular dysfunction and improves 24-hour survival and neurological function in a porcine model of prolonged untreated ventricular fibrillation. Resuscitation. 2011 Dec;82 Suppl 2(0 2):S35-40. doi: 10.1016/S0300-9572(11)70149-6. PMID 22208176
- [Background] Schultz J, Segal N, Kolbeck J, McKnite S, Caldwell E, Yannopoulos D. Sodium nitroprusside enhanced cardiopulmonary resuscitation (SNPeCPR) improves vital organ perfusion pressures and carotid blood flow in a porcine model of cardiac arrest. Resuscitation. 2012 Mar;83(3):374-7. doi: 10.1016/j.resuscitation.2011.07.038. Epub 2011 Aug 22. PMID 21864483
- [Background] Schultz JC, Segal N, Caldwell E, Kolbeck J, McKnite S, Lebedoff N, Zviman M, Aufderheide TP, Yannopoulos D. Sodium nitroprusside-enhanced cardiopulmonary resuscitation improves resuscitation rates after prolonged untreated cardiac arrest in two porcine models. Crit Care Med. 2011 Dec;39(12):2705-10. doi: 10.1097/CCM.0b013e31822668ba. PMID 21725236
- [Background] Yannopoulos D, Matsuura T, Schultz J, Rudser K, Halperin HR, Lurie KG. Sodium nitroprusside enhanced cardiopulmonary resuscitation improves survival with good neurological function in a porcine model of prolonged cardiac arrest. Crit Care Med. 2011 Jun;39(6):1269-74. doi: 10.1097/CCM.0b013e31820ed8a6. PMID 21358401